CLINICAL TRIAL: NCT01993069
Title: Yoga Training for Returning Veterans With Headache
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Bruce Naliboff, PhD, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCC 2013-020286
Record Dates: First submitted 2013-07-16; First posted 2013-11-25 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Post Traumatic Headache; Chronic Daily Headache
MeSH Terms: conditions — Post-Traumatic Headache; Headache Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iyengar-based Yoga Training (Experimental): 6 weekly Iyengar-based yoga classes
  Interventions: Behavioral: Iyengar-based Yoga Training

INTERVENTIONS:
Behavioral: Iyengar-based Yoga Training — 6 weekly Iyengar-based yoga classes

SUMMARY:
The objective of the study is to evaluate the efficacy of a yoga treatment for veterans with mild post-traumatic and chronic tension-type headaches.

Study Aims:

* Does this yoga treatment, targeted toward specific symptoms veterans with mild post-traumatic and chronic tension-type headaches experience, assist in decreasing headaches and associated symptoms?
* Does this yoga treatment, targeted toward specific symptoms veterans with mild post-traumatic and chronic tensions-type headaches experience, assist in improving quality of life?
* Does this yoga treatment, targeted toward specific symptoms veterans with mild post-traumatic and chronic tension-type headaches experience, improve mood?
* Do the effects of yoga on symptoms, mood, and quality of life maintain 2 months post completion of treatment?

DETAILED DESCRIPTION:
The objective of the study is to evaluate the efficacy of a yoga treatment for veterans with mild post-traumatic and chronic tension-type headaches. The yoga will be provided in the form of 6 weekly yoga sessions aimed at providing direct instruction and immediate feedback on postures, breathing, and relaxation techniques in a small group format. The sessions will be led by an experienced yoga instructor who is a part of the study team and have worked with medical patients. A post-yoga 2-month follow-up assessment of self-reported symptoms, mood, and quality of life will also be assessed.

This is a feasibility study to determine if a yoga treatment is received favorably and can be successfully delivered to veterans seeking treatments for post-traumatic and chronic tension-type headaches. This study does not include a comparison group; therefore, we can only make conclusions based on pre to post differences in subjects who participate in the yoga. Our aim for this study is to collect data on the potential benefits of a targeted yoga treatment for symptoms experienced by these subjects, and to then utilize these data to implement a larger study with a comparison group.

ELIGIBILITY:
Inclusion Criteria:

Eligibility determined at screening will be based on the following inclusion criteria: Mild post traumatic headaches or chronic tension-type headaches, diagnosed by a physician. Inclusion criteria also includes the following: 1). Ability to participate in yoga classes (i.e., no physical limitations, mobility issues, or severe chronic medical issues/symptoms such as severe chronic back pain or injury, amputees, being wheelchair bound), 2). Not current involved in regular yoga of more than an hour of yoga per week in a formal setting, 3). If a woman, not currently pregnant or breast feeding, 4). Ages 18 and up (no maximal age limit), 5). Veterans only (no non-veteran populations), and 6). Not currently suffering from severe psychiatric diagnoses (e.g., schizophrenia, bipolar disorder), a history of psychiatric hospitalization, or current substance abuse or dependence.

Exclusion Criteria:

Exclusion based on the following: 1). Age less than 18 years old (not an adult); 2). Not a veteran; 3). Physical limitations, mobility issues, or severe chronic medical issues that may impede one's ability to participate in yoga classes (e.g., wheelchair bound veterans, amputees, those with severe musculoskeletal or nerve pain or injury such as chronic back pain with significantly limited range of motion); 4). Current severe psychiatric diagnoses (e.g., schizophrenia, bipolar disorder) or history of psychiatric hospitalizations; 5). Current substance abuse or dependence; 6). Current regular yoga practice involving more than an hour of yoga per week in a formal setting; and 7). If a woman, currently pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Symptom relief, headache | Post-Treatment, up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Naliboff, PhD, Principal Investigator — University of California, Los Angeles; Milena Zirovich, MD, Principal Investigator — VAGLAHS
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States